CLINICAL TRIAL: NCT07345000
Title: A Randomized, Controlled, Multicenter, Double-blind Phase III Study Evaluating the Efficacy and Safety of Romiplostim N01 Combined With Standard Immunosuppressive Therapy (IST) Versus Placebo Combined With IST in Treatment-naïve Subjects With Severe Aplastic Anemia
Brief Title: A Study of Romiplostim N01 Plus IST vs. Placebo Plus IST for Treatment-Naive Severe Aplastic Anemia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL0911-304
Record Dates: First submitted 2025-12-23; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Treatment-naïve Severe Aplastic Anemia
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Romiplostim N01+ IST (Experimental)
  Interventions: Drug: Romiplostim N01; Drug: Cyclosporine A (CsA); Drug: pALG/ rATG
- Placebo+ IST (Active Comparator)
  Interventions: Drug: Placebo; Drug: Cyclosporine A (CsA); Drug: pALG/ rATG

INTERVENTIONS:
Drug: Romiplostim N01 — Starting from Day 1 of Week 1, administer the initial dose of romiplostim N01: 10 μg/kg. Platelet count (PLT) must be monitored weekly. The dose should be adjusted based on platelet values (adjusted by 5 μg/kg per change, see the table below for specific rules), administered once weekly, with a maximum dose of 20 μg/kg.
  Arms: Romiplostim N01+ IST
Drug: Cyclosporine A (CsA) — Initiate at a dose of 5 mg/kg/day, administered orally in two divided doses (recommended at 12-hour intervals). The dose may be adjusted between 3 and 5 mg/kg/day based on the subject's tolerance.
  Arms: Romiplostim N01+ IST
Drug: pALG/ rATG — 25 mg/kg/day on Days 1 through 5 of Week 1.
  Arms: Romiplostim N01+ IST
Drug: Placebo — Starting from Day 1 of Week 1, administer the initial dose of placebo: 10 μg/kg. Platelet count (PLT) must be monitored weekly. The dose should be adjusted based on platelet values (adjusted by 5 μg/kg per change, see the table below for specific rules), administered once weekly, with a maximum dose of 20 μg/kg.
  Arms: Placebo+ IST
Drug: Cyclosporine A (CsA) — Initiate at a dose of 5 mg/kg/day, administered orally in two divided doses (recommended at 12-hour intervals). The dose may be adjusted between 3 and 5 mg/kg/day based on the subject's tolerance.
  Arms: Placebo+ IST
Drug: pALG/ rATG — 25 mg/kg/day on Days 1 through 5 of Week 1.
  Arms: Placebo+ IST

SUMMARY:
This is a randomized, double-blind, multicenter trial designed to evaluate treatment with romiplostim N01+ IST compared with placebo + IST in the participants with treatment-naïve severe aplastic anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥15 years, regardless of sex (subjects ≥18 years old will be enrolled first; enrollment of subjects aged 15-18 years will commence after sufficient PK/PD data are obtained).
2. Diagnosis of SAA or VSAA according to the British Journal of Haematology (BJH) guidelines. The diagnostic criteria for SAA are as follows:

   ①Bone marrow cellularity <25% of normal; or between 25% and <50%, with residual hematopoietic cells comprising <30%.

   ②Peripheral blood counts must meet at least two of the following three criteria (based on the lowest values from tests within 28 days prior to the first dose):
   1. Absolute neutrophil count (ANC) <0.5×10⁹/L
   2. Platelet count (PLT) <20×10⁹/L
   3. Absolute reticulocyte count (RET) <60×10⁹/L The diagnostic criterion for VSAA is: meeting the SAA criteria + ANC <0.2×10⁹/L.
3. Written informed consent

Exclusion Criteria:

1. History and/or concomitant presence of other primary or secondary bone marrow failure (BMF) syndromes, such as:

   ①Primary: Fanconi anemia, dyskeratosis congenita, congenital amegakaryocytic thrombocytopenia or Shwachman-Diamond syndrome, symptomatic paroxysmal nocturnal hemoglobinuria (PNH), myelodysplastic syndromes (MDS), clonal cytopenia of undetermined significance (CCUS), antibody-mediated BMF, idiopathic cytopenia of undetermined significance (ICUS), etc.
   * Secondary: large granular lymphocyte (LGL) leukemia, infiltration of the bone marrow by other systemic malignancies, myelofibrosis, and acute hematopoietic arrest, etc.

   Note: Asymptomatic PNH and hepatitis-associated SAA may be included if they meet all other inclusion criteria.
2. Evidence of clonal cytogenetic abnormalities at screening.
3. Participation in another clinical trial with investigational drugs or medical devices within 30 days prior to the first dose or within 5 half-lives of the investigational product (whichever is longer).
4. Previous use of any of the following agents prior to the first dose:

   * ATG/ALG

     * Alemtuzumab

       * Mycophenolate mofetil ④Sirolimus

         * Tacrolimus ⑥High-dose cyclophosphamide (≥45 mg/kg/day)
5. Cumulative cyclosporine A (CsA) therapy exceeding 4 weeks prior to the first dose. If cumulative use is ≤4 weeks, a washout period of >14 days prior to the first dose is required.
6. Cumulative use of thrombopoietin receptor agonists (TPO-RAs) for >14 days prior to the first dose, or cumulative use ≤14 days with a washout period of <14 days, including:

   * Romiplostim / Nplate® (romiplostim)

     * Eltrombopag ③Hetrombopag ④Recombinant human thrombopoietin, etc.
7. Previous history of hematopoietic stem cell transplantation.
8. Uncontrolled bleeding and/or infection after standard treatment prior to the first dose [defined as persistent signs/symptoms related to infection without improvement despite appropriate antibiotic and/or other therapy], or requiring intravenous (IV) antibiotic administration.
9. Concomitant active CMV and EBV infection (positive test).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) rate at the 6-month time point of treatment. | During 6 months of therapy
  Proportion of subjects achieving hematopoietic complete response at the 6-month.
  Hematopoietic complete response is defined as: hemoglobin ≥10 g/dL, absolute neutrophil count ≥1×10⁹/L, and platelet count ≥100×10⁹/L.